CLINICAL TRIAL: NCT03943069
Title: Thoracoscopic Bullectomy Versus Thoracoscopic Bullectomy and Pleurodesis For Management of Primary Spontaneous Pneumothorax; A Prospective Multicenter Randomized Controlled Study
Brief Title: Thoracoscopic Bullectomy Versus Thoracoscopic Bullectomy With Pleurodesis in Primary Spontaneous Pneumothorax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: King Fahad Specialist Hospital Dammam (Other); Qatif Central Hospital (Other); Johns Hopkins Aramco Healthcare (Other)
Responsible Party: Principal Investigator, Hatem Elbawab, Associate professor, Imam Abdulrahman Bin Faisal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThorSurg_2014-04
Record Dates: First submitted 2019-04-19; First posted 2019-05-09 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Thoracic Surgical Procedures
MeSH Terms: interventions — Pleurodesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with PSP (Experimental): Patient who will be admitted with primary spontaneous pneumothorax.
  Interventions: Procedure: Thoracoscopic bullectomy alone; Procedure: Thoracoscopic bullectomy with pleurodesis

INTERVENTIONS:
Procedure: Thoracoscopic bullectomy alone — Thoracoscopic stapling of emphysematous like changes (ELCs) to control the air leak from the lung bullae.
  Other Names: VATS Bullectomy
Procedure: Thoracoscopic bullectomy with pleurodesis — Thoracoscopic stapling of emphysematous like changes (ELCs) to control the air leak from the lung bullae.in addition to mechanical pleurodesis.
  Other Names: VATS Bullectomy with pleurodesis

SUMMARY:
The exact pathogenesis of PSP is controversial. A few theories has been proposed contributing to the pathogenesity of the PSP as emphysematous like changes (ELCs) which lead to the formation and rupture of the lung bullae or blebs; and increased pleural porosity which is an abnormality of the visceral pleura. The Video-Assisted Thoracoscopic Surgery with bullectomy only is an effective preventive method of PSP recurrence. Adding mechanical pleurodesis to bullectomy is still questionable in the literature. This prospective multicenter study will identify the rate of PSP recurrence after thoracoscopic bullectomy only versus thoracoscopic bullectomy with mechanical pleurodesis.

DETAILED DESCRIPTION:
Background The pneumothorax may be defined as presence of air in the pleural cavity which then leads to a decrease in lung expansion, and consequently lung collapse. The pneumothorax occurs due to air lodged at the pleural space either between the pleural cavity and the alveolar between the pleural cavity and the atmosphere; or the presence of organisms that produce gases (1).

The pneumothorax can be classified into spontaneous or traumatic. The spontaneous pneumothorax (SP) is either classified into primary SP that has no underlying lung disease; or secondary SP that occurs in underlying lung disease as Chronic Obstructive Pulmonary Diseases (COPDs), or in conjugation with menstrual period causing catamenial pneumothorax (1).

The exact pathogenesis of primary spontaneous pneumothorax (PSP) is controversial. The theories beyond the pathology of PSP has includes: emphysematous like changes (ELCs) which cause formation and rupture of the blebs or bullae; increased pleural porosity which is an abnormality of the visceral pleura seen under fluorescein lighting; and inflammation of the distal airways which lead to fibrotic change and compensatory emphysematous bulla (2). The development of the previous etiologies are linked to genetic predisposition, anatomical abnormalities, connective tissues abnormalities, body mass index under 18.5 kg/m2, decrease caloric intake, and apical ischemia(3).

In the literature there was a superiority in treatment of PSP with the Video-assisted thoracoscopic surgery (VATS) is in compare to thoracotomy, as it has less tissue damage, less postoperative pain, less hospitalization stay, better cosmetic outcome, and earlier return to normal daily life activities (4). The debate on the ideal preventive method of PSP recurrence using VATS spotlights on the main etiologies of the treatment of bleb and bullae by the bullectomy and the pleural abnormalities by pleurodesis(5).

VATS with bullectomy alone is an effective method of decreasing the chance of PSP recurrence, while additive of mechanical pleurodesis is questionable as different studies showed variable results(6-8). This multicenter randomized control trial study will compare the recurrence rate of PSP post thoracoscopic bullectomy alone in compare with thoracoscopic bullectomy in addition to mechanical pleurodesis.

Methodology Study setting This is a randomized control trial study which will be held at the following hospitals: King Fahad Hospital of University (KFHU), Qatif Central Hospital (QCH), King Fahad Specialist Hospital Dammam (KFSH), and John Hopkins Aramco Healthcare.

The Study will include all Saudi and non-Saudi patients, male or female, age between 16-45-year-old, diagnosed with PSP. The exclusion criteria: any patient with previous thorax surgery history, patient undergoing thoracotomy and patient with hemothorax.

Sample Size In order to calculate the sample size, the recurrence rate of the Thoracoscopic Bullectomy and Mechanical Pleurodesis (TB+MP) was conservatively estimated to be lower than 2%, whilst the recurrence rate of the Thoracoscopic Bullectomy (TB) group was estimated to be 12%. To attain a study power of 80% with an alpha error of 0.05 the sample size was estimated to be 202. Assuming a 15% loss to follow-up rate, at least 232 subjects between groups will be selected.

Randomization and Masking Computer generated randomization will be used, and to ensure random allocation and concealment, surgeons from the multiple centers that have been included will contact a central randomization service provided by a distant and blinded research fellow not involved in treatments upon arrival of patients who fulfill the inclusion criteria that have been set a priori to either the TB group or the Thoracoscopic TB+MP group.

Surgical technique The patients will be operated under general anesthesia with ventilation of one lung using double-lumen endotracheal tube.

Two or three ports thoracoscopic technique will be used to open and visualize the thoracic cavity. The procedure whether bullectomy alone or bullectomy with pleurodesis will be selected randomly preoperatively after informed consent. Wedge resection using an endoscopic stapler will target the bullae. In addition to the bullectomy the investigators will do mechanical pleurodesis according to the randomization by pleural abrasion, and consistent techniques for pleural abrasion the investigators will maintain with regard to the extent and aggressiveness of abrasion. In the mechanical pleurodesis, the mesothelial layer of the parietal pleura will be abraded from the cupola of the thoracic cavity apex to the 5th intercostal space.

Post-operatively a traditional chest drainage system will be connected to the patient's chest for monitoring the air-leak and fluid drainage. The traditional chest drainage consists of drainage chamber, water-seal chamber, and suction control.

Data Collection Medical records; chest x-ray or Computed Tomographic Scan (CT-scan) result; presenting symptoms; operative time; intraoperative blood loss; postoperative thoracic drainage amount, air-leakage duration, chest tube duration and pain scale score; length of hospital stay; and details of follow-up will be assessed by the same treating inverstigator.

All patients will be followed-up in one week, one months, three months and six months looking for pneumothorax recurrence. Nevertheless, patients will be instructed to return to the emergency department if they develop chest pain, shortness of breath, or if symptoms are suggestive of pneumothorax recurrence. All recurrence cases will be confirmed by chest X-ray or CT-scan.

Statistical analysis STATA Statistical Software version 15 will be used for data analysis. Analyses will commence with a description of the population where percentages and means along with their respective standard deviations will be reported. Multi-variate analyses will be based on the intention-to-treat principle. All tests of significance will be 2-sided. A comparison will be made between the two treatment groups based on the amount of drainage in (ml) using the hazard ratio and its respective confidence interval which will be calculated from a Cox proportional hazards model. All outcome measures will be adjusted for age, sex, smoking index, BMI, and physical activity. A p-value of less than 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Primary spontaneous pneumothorax
* Male or female
* Age 16-45

Exclusion Criteria:

* Hemopneumothorax
* Previous thoracic surgical intervention
* Patient undergoing thoracotomy

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 232 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-11-25 (Estimated); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pneumothorax | 6 months
  The evaluation of recurrence of primary spontaneous pneumothorax will be via the radiological studies (Chest x-ray) that will be performed during the follow-up visits in 1 week, 1 month, 3 months and 6 months after hospital discharge. Moreover, symptoms such as respiratory distress and ipsilateral chest pain during the follow up period will be considered as a recurrence of pneumothorax which requires further evaluation and confirmation by radiological studies. The number of recurrences during the follow up period will be compared between the two groups for any statistical difference.

SECONDARY OUTCOMES:
Drainage and air leak | 1 week
  The amount and characteristics of chest tube drainage and the degree and duration of air-leak during hospital stay will be recorded. The results will be compared between both groups and will be evaluated for any statistical difference.
Postoperative Pain | 1 week
  Visual analogue scales (VAS) will assess the pain for each patient from the first day postoperative till date of hospital discharge. The scale will be used to describe the pain severity from 0 to 10. The 0 score is considered as no pain, the 5 score is considered as distressing pain, and the score at 10 is considered as the most severe pain. The result will be compared between both groups and will be evaluated for statistical difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years

REFERENCES:
- [Background] Noppen M, De Keukeleire T. Pneumothorax. Respiration. 2008;76(2):121-7. doi: 10.1159/000135932. Epub 2008 Jun 26. PMID 18708734
- [Background] Grundy S, Bentley A, Tschopp JM. Primary spontaneous pneumothorax: a diffuse disease of the pleura. Respiration. 2012;83(3):185-9. doi: 10.1159/000335993. Epub 2012 Feb 15. PMID 22343477
- [Background] Noppen M. Spontaneous pneumothorax: epidemiology, pathophysiology and cause. Eur Respir Rev. 2010 Sep;19(117):217-9. doi: 10.1183/09059180.00005310. PMID 20956196
- [Background] Huh U, Kim YD, Cho JS, I H, Lee JG, Lee JH. The Effect of Thoracoscopic Pleurodesis in Primary Spontaneous Pneumothorax: Apical Parietal Pleurectomy versus Pleural Abrasion. Korean J Thorac Cardiovasc Surg. 2012 Oct;45(5):316-9. doi: 10.5090/kjtcs.2012.45.5.316. Epub 2012 Oct 9. PMID 23130305
- [Background] Noppen M, Baumann MH. Pathogenesis and treatment of primary spontaneous pneumothorax: an overview. Respiration. 2003 Jul-Aug;70(4):431-8. doi: 10.1159/000072911. PMID 14512683
- [Background] Alayouty HD, Hasan TM, Alhadad ZA, Omar Barabba R. Mechanical versus chemical pleurodesis for management of primary spontaneous pneumothorax evaluated with thoracic echography. Interact Cardiovasc Thorac Surg. 2011 Nov;13(5):475-9. doi: 10.1510/icvts.2011.270280. Epub 2011 Aug 9. PMID 21828109
- [Result] Zhang Z, Du L, Feng H, Liang C, Liu D. Pleural abrasion should not routinely preferred in treatment of primary spontaneous pneumothorax. J Thorac Dis. 2017 Apr;9(4):1119-1125. doi: 10.21037/jtd.2017.03.124. PMID 28523168
- [Result] Horio H, Nomori H, Kobayashi R, Naruke T, Suemasu K. Impact of additional pleurodesis in video-assisted thoracoscopic bullectomy for primary spontaneous pneumothorax. Surg Endosc. 2002 Apr;16(4):630-4. doi: 10.1007/s00464-001-8232-5. Epub 2002 Jan 9. PMID 11972203